CLINICAL TRIAL: NCT01948856
Title: CLEARI (Clinical Efficacy Assessment on Recurrent Upper-Respiratory Tract Infections) Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pierre Fabre Medicament (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: J0022X ST 3 02; 2013-001760-31 (EudraCT Number)
Record Dates: First submitted 2013-09-19; First posted 2013-09-24 (Estimated); Last update posted 2017-02-03 (Estimated); Status verified 2017-02

CONDITIONS: Recurrent Upper-Respiratory Tract Infections
Keywords: Recurrent common cold; laryngitis; pharyngitis/tonsillitis; acute rhinitis; acute rhinosinusitis; acute otitis media
MeSH Terms: conditions — Respiratory Tract Infections; Common Cold; Laryngitis; Pharyngitis; Tonsillitis; Otitis Media

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- J022X ST (Experimental)
  Interventions: Drug: J022X ST
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: J022X ST — Oral administration - During 6 months and according to the approved summary of product characteristics : 1 sachet per day in the morning on an empty stomach
  * First month: 4 consecutive days per week during 3 consecutive weeks
  * 5 next months: 4 consecutive days per month at monthly intervals
  Arms: J022X ST
Drug: Placebo — Oral administration - During 6 months : 1 sachet per day in the morning on an empty stomach
  * First month: 4 consecutive days per week during 3 consecutive weeks
  * 5 next months: 4 consecutive days per month at monthly intervals
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the efficacy and safety of J022X ST for prevention of Recurrent Upper-Respiratory Tract Infections (RURTI) compared to placebo in children of younger age who develop infectious diseases more frequently than other children of this age in general.

ELIGIBILITY:
Key Inclusion Criteria:

Patients with all the following criteria will be eligible for inclusion in Year 1:

* Children, male or female
* Aged 3 to 4 years
* Children known for recurrent URTIs in the past year (based on medical recording or reported history)
* Children at risk for URTI in the physician's opinion (e.g. absence of breastfeeding, hospitalization in the previous year, tonsillectomy or adenoidectomy, parental smoking, daycare institution or nursery school, early schooling, prematurity, low weight at birth, malnutrition, failure to thrive).

Patients with all the following criteria will be eligible for randomisation in Year 2:

* Children, male or female
* Aged 4 to 5 years
* Suffering from RURTI, i.e. at least 6 URTI episodes medically confirmed, with a maximum of 18, during the Year 1 of the study.

Key Exclusion Criteria:

Presence of diseases (Chronic suppurative otitis media, acute broncho-pulmonary infection, Immune deficiency or disorders, surgery of respiratory tract, cystic fibrosis…) or treatments (chronic use of corticosteroids, bronchodilators, ...) that may impact the safety, the interpretation of the results and/or the participation of the subject in the study

Ages: 3 Years to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1003 (Actual)
Dates: Start 2013-09; Primary Completion 2016-10-17 (Actual); Study Completion 2016-12-13 (Actual)

PRIMARY OUTCOMES:
Number of Upper-Respiratory Tract Infections (URTI) episodes medically assessed over year 2 | at each infectious episode over year 2
  Each URTI episodes will be medically assessed by the investigator by a thorough medical examination.

CONTACTS AND LOCATIONS:
Overall Officials: Karim KEDDAD, MD, Study Director — Pierre Fabre Medicament
Locations (24):
- Italy (7):
  - Ancona
  - L’Aquila
  - Milan
  - Modena
  - Napoli
  - Roma
  - Varese
- Lithuania (3):
  - Kaunas
  - Panevezys
  - Vilnius
- Poland (6):
  - Lesznowola
  - Lublin
  - Ostrołęka
  - Warsaw
  - Węgrów
  - Wołomin
- Romania (6):
  - Bacau
  - Brasov
  - Bucharest
  - Constanța
  - Craiova
  - Sibiu
- Russia (2):
  - Moscow
  - Saint Petersburg